CLINICAL TRIAL: NCT05503875
Title: Immunoclassification of Psoriasis: a Strategy for Precision Medicine
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0205
Record Dates: First submitted 2022-07-11; First posted 2022-08-17 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Immunoclassification; Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; secukinumab; ixekizumab; guselkumab; Janus Kinase Inhibitors; Methotrexate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): Patients will be treated with adalimumab, secukinumab, ixekizumab, guselkumab, Jak inhibitors or methotrexate.
  Interventions: Biological: adalimumab, secukinumab, ixekizumab, guselkumab, Jak inhibitors, methotrexate

INTERVENTIONS:
Biological: adalimumab, secukinumab, ixekizumab, guselkumab, Jak inhibitors, methotrexate — Psoriasis patients will be treated with adalimumab, secukinumab, ixekizumab, guselkumab, Jak inhibitors or methotrexate.

SUMMARY:
Through the combination of clinical manifestations and omics, the investigators aim to explore the skin cell atlas in different stages of psoriasis lesions, establish a clinical classification standard for psoriasis, and guide the precise treatment of psoriasis.

DETAILED DESCRIPTION:
Psoriasis is a heterogeneous condition that can affect skin and other structures. Over the past decade, considerable advances have been made both in our understanding of the pathogenesis of psoriasis and in the revolutionized immunotherapy of its diverse manifestations. Psoriasis heterogeneity and its cutaneous microenvironment is the leading cause of resistance in patients.

Novel approaches, including single-cell RNA sequencing technology and CyTOF, are proposed as methodological solutions. By their combination with immunotherapy, we can specifically evaluate the mechanism of psoriasis in the face of immunotherapy agents at the single-cell resolution by detecting the transcriptional activity of cytokines, immune checkpoints, screening neoantigens with high transcription levels, identifying rare cells, and assisting the dissection of the critical immune-metabolic pathways in this complex disease. We aim to improve short-term and long-term precision treatment strategies for patients with psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1.18 to 75 years of age 2.Moderate to severe chronic psoriasis, BSA≥3% 3.Duration of psoriasis≥6 months 4.Patients must be candidate for systemic therapy 5.Informed consent must be obtained 6.For female, ß-hCG test is negative and contraception is accepted

Exclusion Criteria:

1. Having severe infections, including hepatitis, HIV and tuberculosis
2. Having significant allergies to biological agents
3. Having a history of malignancy
4. Refusal of contraception
5. Having serious or unstable/uncontrolled illnesses

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in the number of immune cells (dendritic cells, macrophages) in the lesional skin, non-lesional skin of psoriasis patients and healthy skin. | 16 months
  The intensity of specific cell subsets will be assessed by flow cytometry in psoriasis patients and healthy controls.
Molecular analysis of psoriasis lesional skin by single-cell RNA sequencing. | 16 months
  To analyze the intensity of cytokines or chemokines, such as IL-17, IL-23, TNF in the dermis and epidermis of psoriasis patients

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No